CLINICAL TRIAL: NCT04862689
Title: A Prospective, Multicenter, Single-arm Investigation of the Ringer Perfusion Balloon Catheter (Ringer PTCA Study)
Brief Title: Investigation of the Ringer Perfusion Balloon Catheter (Ringer PTCA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Solutions LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST3170
Record Dates: First submitted 2021-04-12; First posted 2021-04-28 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-04

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental (Experimental): Adult subjects clinically indicated for non-emergent percutaneous coronary intervention (PCI) as a stand-alone procedure or following non-emergent diagnostic angiography performed during the same procedure that, in the physician's estimation, requires prolonged balloon inflation with distal perfusion.
  Interventions: Device: Ringer Perfusion Balloon Catheter

INTERVENTIONS:
Device: Ringer Perfusion Balloon Catheter — Non-emergent Percutaneous Coronary Intervention (PCI) for treatment of a coronary artery lesion with Ringer Perfusion Balloon Catheter.

SUMMARY:
The objective of this study is to demonstrate safe and effective use of the Ringer perfusion balloon catheter for dilatation/pre-dilatation of coronary stenoses during percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm clinical study. The study will be conducted in 3 to 5 investigational sites in the US and Canada and will enroll up to 60 participants. The population for this study is adult participants undergoing non-emergent percutaneous coronary intervention (PCI) as a stand-alone procedure or following non-emergent diagnostic angiography performed during the same procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects >18 years old.
* Patients undergoing clinically indicated non-emergent PCI as a stand-alone procedure or in combination with diagnostic angiography during the same procedure.
* Study target lesion characteristics: a) native de-novo coronary stenosis of at least 70% visually estimated stenosis, or at least 50% visually estimated stenosis and shown to be physiologically significant by flow-mediated criteria (FFR <0.80, IFR <0.91); b) estimated reference vessel diameter 2.0-4.5mm; c) lesion length <25mm; d) calcification not greater than mild.
* Per investigator assessment, the patient may benefit from inflation distal perfusion during balloon inflation. Examples include, but are not limited to: (i) LV systolic dysfunction with LVEF<50% by any modality; (ii) a territory subtended by the target vessel downstream from the target lesion that is estimated to be in excess of 25% of viable LV mass; (iii) prior hemodynamic or electrical instablility during intervention on the target lesion; (iv) the potential to avoid placement of a coronary stent if a stent-like result can be achieved through prolonged balloon inflation.
* Female subjects of childbearing potential must have a negative pregnancy test per standard of care for PCI and be practicing contraception.
* Informed consent provided.

Exclusion Criteria:

* Hemodynamic or arrhythmic instability within 48 hours or a myocardial infarction within 72 hours of PCI.
* More than 2 lesions planned during index PCI.
* Procedural complication developing prior to PCI of study target.
* Ejection fraction (EF) <25%.
* Creatinine clearance (Cr-Cl) <25 mg/dL.
* Baseline flow at study target <TIMI-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of device success in dilatation/pre-dilatation of coronary stenosis during PCI. | During Procedure
  Successful delivery, inflation, deflation and withdrawal of the Ringer device; final thrombolysis in myocardial infarction (TIMI) flow grade of 3 at the conclusion of the PCI procedure.
Rate of clinically relevant events | Discharge or 30 days, whichever comes first
  Rate of Ringer related complications arising during delivery, inflation or removal of Ringer; freedom from major cardiac adverse events (MACE)

SECONDARY OUTCOMES:
Successful PCI | During Procedure
  Final residual stenosis ≤20% diameter stenosis (in-stent) or ≤50% diameter stenosis (stand-alone balloon) by visual angiographic estimation and freedom from MACE.
TIMI Flow | During Procedure
  Maintenance of TIMI-2 or -3 flow into distal coronary bed during Ringer inflation
Ringer Inflation | During Procedure
  Tolerance of at least one Ringer inflation greater than one minute (prolonged inflation) at target site (measured with symptoms, ECG, hemodynamics).

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Lane, Study Director — Teleflex; Kathleen Kearney, MD, Principal Investigator — University of Washington
Locations (7):
- United States (4):
  - Torrance Memorial Medical Center, Torrance, California
  - Brigham & Women's Hospital, Boston, Massachusetts
  - St. Luke's Hospital, Kansas City, Missouri
  - University of Washington Medical Center, Seattle, Washington
- Canada (3):
  - Heart Health Institute, Scarborough Village, Ontario
  - Sunnybrook Heath Sciences Center, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No